CLINICAL TRIAL: NCT02398123
Title: Transversus Abdominis Plane (TAP) Blocks Versus Caudal Block for Postoperative Pain Control After Unilateral Lower Abdominal Surgeries in Pediatrics: A Prospective, Randomized Study.
Brief Title: Transversus Abdominis Plane Versus Caudal Block for Pediatrics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUH-Feb-2015
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Lower Abdominal Surgery
Keywords: Transversus Abdominis Plane; caudal block; postoperative pain; children
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transversus abdominis plane block (Active Comparator): Transversus Abdominis Plane block
  Interventions: Other: Transversus abdominis plane block; Drug: Bupivacaine
- Caudal block (Placebo Comparator): Caudal block
  Interventions: Other: Caudal block; Drug: Bupivacaine

INTERVENTIONS:
Other: Transversus abdominis plane block — Children who received transversus aAbdominis plane block with 0.25% bupivacaine with epinephrine 1 mL/kg guided by ultrasound
  Arms: Transversus abdominis plane block
Other: Caudal block — Children who received caudal 0.25% bupivacaine 1 mL/kg
  Arms: Caudal block
Drug: Bupivacaine

SUMMARY:
The transversus abdominis plane (TAP) block is a relatively simple technique that provides myocutaneous anesthesia that, as part of a multimodal analgesic treatment, may be useful in the prevention and treatment of parietal postoperative pain.

Initial experience with ultrasound TAP block demonstrated efficacy of the echo guided technique in different surgical procedures such as cesarean section, appendicectomy, laparoscopic cholecystectomy, infra umbilical surgery in adult and pediatric patients. Recently published clinical trials suggest that TAP block may represents an effective alternative to epidural anesthesia but further studies in larger population are necessary.

Transversus-abdominis plane (TAP) block was found to increase analgesic consumption low thoracic-epidural analgesia (TEA) in ischemic heart disease patients after abdominal laparotomy (2). Others found comparable results between continuous transversus abdominis plane technique and epidural analgesia in regard to pain, analgesic use and satisfaction after abdominal surgery(3). The TAP block affords effective analgesia with opioid sparing effects, technical simplicity, and long duration of action. Some disadvantages include the need for bilateral block for midline incisions and absence of effectiveness for visceral pain (4). TAP block has been associated with good pain relief and decreased intraoperative and postoperative opioids requirements after laparoscopic surgery (5). The analgesic efficacy of the TAP block has been demonstrated in prospective randomized trials compared with placebo, in different surgical procedures such as abdominal surgery, hysterectomy, retro pubic prostatectomy, Caesarean section, laparoscopic cholecystectomy, and appendicectomy (6, 7, 8, 9, 5 and 10 respectively). All these studies have reported superiority of the TAP block in terms of reduction in visual analogue scale scores and morphine consumption. In this study the investigators try to compare Transversus Abdominis Plane (TAP) blocks versus caudal block for postoperative pain control after lower abdominal surgeries in pediatrics.

DETAILED DESCRIPTION:
Children aged 1-7 years undergoing lower abdominal surgeries would be recruited in this randomized study.

Children would be monitored by electrocardiogram, pulse oximeter and non-invasive blood pressure.

After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 33% oxygen and 66% nitrous oxide; 1ug/kg fentanyl is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory (jaw relaxed, lash reflex disappeared, no coughing, gagging, swallowing).

Anesthesia would be maintained with 2% sevoflurane and nitrous oxide.

An increase in blood pressure or heart rate by more than 15% from preoperative value was defined as insufficient analgesia and was treated with fentanyl 0.5 µ/kg. Saline dextrose5% (1:1) solution was infused in a dose of 12 ml/ kg /h.

Children were transferred from PACU to day-surgery unit (DSU) if they achieved Modified Aldrete Score of ten.

Patients received rectal paracetamol 15 mg/ kg every 6 hours. Tramadol 1mg/kg is rescue analgesic.

ELIGIBILITY:
Inclusion Criteria:

* Children
* Lower abdominal surgery

Exclusion Criteria:

* Allergy to study medications
* Contraindications to caudal block
* Contraindications to transversus abdominis block

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time for first analgesic request | 24 hours after surgery
  By investigators until hospital discharge, then through telephone interview with parents after that

SECONDARY OUTCOMES:
Total opioid consumption | 24 hours after surgery
  By investigators until hospital discharge, then through telephone interview with parents after that
Sedation level | 12 hours after surgery
  Sedation level would be evaluated using a four-point sedation scale, 0=eyes open spontaneously, 1=eyes open to speech, 2=eyes open when shaken, 3=un arousable.
Parent satisfaction scores | 24 hours after surgery
  By investigators until hospital discharge, then through telephone interview with parents after that
Modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS), | 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 18 h, 24 h after surgery
  By investigators until hospital discharge, then through telephone interview with parents after that

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Eldeeb, MD, Study Chair — Associate Professor of Anesthesia and Surgical ICU, Mansoura University , Mansoura City, Egypt
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt